CLINICAL TRIAL: NCT02060916
Title: Study to Evaluate the Safety and Efficacy of PAZ320 When Added to Oral Agents or Insulin in Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Evaluate the Safety and Efficacy of PAZ320 in Patients With Type 2 Diabetes
Acronym: PAZ320
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PAZ320-002
Record Dates: First submitted 2013-11-18; First posted 2014-02-12 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Treated With Insulin
MeSH Terms: interventions — PAZ320

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- PAZ320 (Experimental): Patients will all take part in the control arm of the study and then be crossed over into treatment with PAZ320 at two different dosages.
  Interventions: Drug: PAZ320

INTERVENTIONS:
Drug: PAZ320 — Single-center pilot study, open label dose escalation design

SUMMARY:
This study is to evaluate the effect that PAZ320 has on post-prandial glucose excursions measured via continuous glucose monitoring and its adverse effect profile in humans.

DETAILED DESCRIPTION:
In this study, the investigators seek to evaluate the effect that PAZ320 has on post-prandial glucose excursions measured via continuous glucose monitoring and its adverse effect profile in humans. Continuous glucose monitors (CGM) are minimally invasive devices that measure glucose levels in interstitial fluid. A small wire is inserted subcutaneously which transmits the ambient subcutaneous glucose concentration every 5 minutes to a wireless recorder. In usual use, the patient can see these data and graph the previous 1, 3 or 9 hours to identify trends or look back over time (ie over night). In our study, the patient will be blinded to the data so as not to confound results, as it has been noted in another study that patient's blood sugar control was better when they were able to see CGM results and modified their diet. CGM's have been shown to have clinical accuracies of 95.5-98.9% and have been used in clinical trials and found to be safe. Having the patient do a finger-stick glucose intermittently during the time they are wearing the CGM improves accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18-75 years;
* Subjects diagnosed with Type 2 Diabetes mellitus;
* Subjects currently on oral agents or insulin;
* Body mass index 25 to 40 kg/m2;
* Subjects able to comply with study procedures and sign informed consent
* A1c less than or equal to 9%

Exclusion Criteria:

* Medication (other than diabetes medications or insulin) or dietary supplement known to affect glucose or galactose metabolism
* Use of acetaminophen-containing products
* Lactose or galactose intolerance
* History of eating disorder
* Food allergy or severe food intolerance
* Pregnant or lactating female
* Subjects with diabetes mellitus treated with very high dose of sulfonylureas (glyburide>20 mg/day, , glimepiride >8 mg per day, and glipizide >20 mg per day) α-glucosidase inhibitors (acarbose ), or meglitinides (repaglinide >6 mg per day)), ;
* Subject with gastrointestinal disease that may interfere with absorption of the investigational products at discretion of investigator, including but are not limited to malabsorption syndromes and gastric ulcer;
* Subject has received any investigational agent within 30 days prior to the first dose of investigational product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of the food supplement PAZ320 on post-prandial glucose excursion | 1 week

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Trask, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Jefferson, New Hampshire, United States